CLINICAL TRIAL: NCT04025632
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Efficacy of Zilucoplan in Subjects With Immune-Mediated Necrotizing Myopathy
Brief Title: Safety and Efficacy Study of Zilucoplan in Subjects With Immune-Mediated Necrotizing Myopathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated based on the primary efficacy endpoint analysis after the first data lock.
Sponsor: Ra Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RA101495-02.202
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Results first posted 2022-05-16 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Immune Mediated Necrotizing Myopathy
MeSH Terms: interventions — zilucoplan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 0.3 mg/kg zilucoplan (Experimental): Daily subcutaneous (SC) injection
  Interventions: Drug: zilucoplan
- Placebo (Placebo Comparator): Daily subcutaneous (SC) injection
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: zilucoplan — Daily subcutaneous (SC) inection
  Arms: 0.3 mg/kg zilucoplan
Other: Placebo — Daily subcutaneous (SC) inection
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of zilucoplan in patients with Immune-Mediated Necrotizing Myopathy (IMNM). Subjects will be randomized in a 1:1 ratio to receive daily SC doses of 0.3 mg/kg zilucoplan or matching placebo for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of IMNM (Immune-Mediated Necrotizing Myopathy)
* Positive serology for anti-3-hydroxy-3-methyl-glutaryl-coenzyme A reductase (HMGCR) or anti-signal recognition particle (SRP) autoantibodies
* Clinical evidence of weakness (≤ grade 4 out of 5) on manual muscle testing in at least one proximal limb muscle group
* Creatine kinase (CK) of >1000 U/L at Screening
* No change in corticosteroid dose for at least 30 days prior to Baseline or anticipated to occur during the first 8-weeks on study
* No changes in immunosuppressive therapy, including dose, for at least 30 days prior to Baseline or anticipated to occur during the first 8-weeks on study

Exclusion Criteria:

* History of meningococcal disease
* Current or recent systemic infection within 2 weeks prior to Screening or infection requiring intravenous (IV) antibiotics within 4 weeks prior to Screening
* Recent initiation of intravenous immunoglobulin (IVIG) (i.e., first cycle administered less than 90 days prior to Baseline)
* Rituximab use within 90 days prior to Baseline or anticipated to occur during study
* Statin use within 30 days prior to Baseline or anticipated to occur during study
* Plasma exchange within 4 weeks prior to Baseline or expected to occur during the 8-week Treatment Period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — UCB Pharma
Locations (18):
- United States (14):
  - University of California Los Angeles, Los Angeles, California
  - University of California Irvine, Orange, California
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - National Institute of Health, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University School of Medicine in Saint Louis, St Louis, Missouri
  - Northwell Health Neuroscience Institute, Great Neck, New York
  - The Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Wesley Neurology Clinic, Memphis, Tennessee
  - Austin Neuromuscular Center, Austin, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
- Hôpital Universitaire Pitié Salpêtrière, Paris, France
- Amsterdam UMC, Amsterdam, Netherlands
- United Kingdom (2):
  - University College London Hospitals NHS Foundation Trust, London
  - Salford Royal NHS Barnes Clinical Research Facility, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was performed in 4 countries (France, the Netherlands, the United Kingdom, and the United States of America) between 07 November 2019 and 14 June 2021.
Pre-assignment Details: Of the 37 participants who were screened, 10 participants were deemed ineligible and were screen failures. 27 participants with immune-mediated necrotizing myopathy were randomized in a 1:1 ratio to receive zilucoplan 0.3 mg/kg or a matching placebo for the 8-week Treatment Period in the Main Portion of the study. All eligible participants were given the option to receive daily subcutaneous (SC) zilucoplan 0.3 mg/kg in the Extension Portion of the study.
Groups:
- Placebo: Participants were randomized to receive daily SC doses of matching placebo during the 8-week Main Portion of the study. All eligible participants were given the option to receive daily SC zilucoplan 0.3 mg/kg in the Extension Portion of the study.
- Zilucoplan 0.3 mg/kg: Participants were randomized to receive daily SC doses of zilucoplan 0.3 mg/kg during the 8-week Main Portion of the study. All eligible participants were given the option to receive daily SC zilucoplan 0.3 mg/kg in the Extension Portion of the study.
Period: Overall Study
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
Started | 15 | 12
Completed Main Portion | 15 | 12
Started Main Portion Safety Follow-up (Refers to study participants who completed the 8-week blinded treatment period in the Main Portion of the study and had not entered the Extension Portion.) | 2 | 0
Completed Main Portion Safety Follow-up (Refers to study participants who completed the 8-week blinded treatment period in the Main Portion of the study and had not entered the Extension Portion.) | 0 | 0
Started Extension Portion | 13 | 12
Completed (Completed Main Portion, Main Portion Safety Follow-up or Extension Portion.) | 0 | 0
Not Completed | 15 | 12
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Study Terminated by Sponsor | 10 | 9
Not completed — Physician Decision | 3 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg | Total
Number analyzed (Participants) | 15 | 12 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (13.6) | 56.9 (9.0) | 54.6 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 8 | 5 | 13
  Unknown or Not Reported | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  White | 10 | 7 | 17
  Other/Mixed | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
  Missing | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline to Week 8 in Serum Creatine Kinase (CK) Levels
Description: All laboratory samples were obtained prior to administration of study drug at applicable visits. CK levels were measured by a central laboratory.
Time Frame: Baseline (Day 1) and end of Main Portion (Week 8)
Population: The ITT Population with no missing observations at Baseline and Week 8.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 14 | 10
percentage change | -20.72 (31.22) | -9.86 (26.06)
Statistical Analysis 1: Comparison: Placebo vs Zilucoplan 0.3 mg/kg; Test type: Superiority; p = 0.464, 2-sided Van Elteren test — Conducted using a 2-sided Van Elteren test, which represents an extension of the Wilcoxon rank sum test for comparing 2 treatments in a stratified experiment using within-stratum ranks assigning greater weight to rank sums from smaller strata; Wilcoxon-Mann-Whitney odds = 0.55, 95% CI 2-sided [0.19 to 1.57] — The magnitude of association between treatment groups was expressed as in Wilcoxon-Mann-Whitney odds followed by the 95% confidence intervals

2. Primary Outcome: Number of Participants Who Experienced a Treatment-Emergent Adverse Event (TEAE)
Description: A TEAE was defined as:
  * An adverse event (AE) that occurred after study treatment start that was not present at the time of treatment start.
  * An AE that increased in severity after treatment start if the event was present at the time of treatment start.
Time Frame: Baseline (Day 1) to end of Main Portion (Week 8)
Population: The Safety Population included all participants who have received at least 1 dose of study drug, with participants analyzed based on the actual study treatment received.
Measure: Count of Participants; unit: Participants
Groups:
- Main Portion: Placebo: Participants were randomized to receive daily SC doses of matching placebo during the 8-week Main Portion of the study.
- Main Portion: Zilucoplan 0.3 mg/kg: Participants were randomized to receive daily SC doses of zilucoplan 0.3 mg/kg during the 8-week Main Portion of the study.
Arm/Group | Main Portion: Placebo | Main Portion: Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 15 | 12
Participants | 13 | 9

3. Secondary Outcome: Number of Participants Who Achieve at Least Minimal Response Based on the American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Response Criteria Scale
Description: The ACR/EULAR scale utilized a conjoint analysis-based continuous model using absolute percent change from Baseline in core set measures (physician, patient, and Myositis Disease Activity Assessment Tool (MDAAT); muscle strength; Health Assessment Questionnaire (HAQ); and muscle enzyme levels). A total improvement score (range 0-100) was determined by summing scores for each core set measure and comparing improvement in each respective core set measure. The threshold for minimal improvement was ≥20 in the total improvement score with higher scores indicating a better outcome.
Time Frame: Baseline (Day 1) and end of Main Portion (Week 8)
Population: The ITT Population with no missing observations at Baseline and Week 8.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 14 | 11
Participants | 7 | 6
Statistical Analysis 1: Comparison: Placebo vs Zilucoplan 0.3 mg/kg; Test type: Superiority; p = 0.919, Regression, Logistic — P-value for the comparison of treatment groups was calculated using logistic regression with investigational medicinal product and strata as fixed factors; Odds Ratio (OR) = 1.088, 95% CI 2-sided [0.214 to 5.535]

4. Secondary Outcome: Change From Baseline to Week 8 in Triple Timed Up and Go Test (3TUG) Time
Description: The 3TUG test involved the ambulatory participant getting up from a seated position in a chair, walking at their normal pace for 3 meters, turning around, walking back to the chair, and sitting down. This sequence was repeated 3 times without rest, and the 3TUG test time is the average of the 3 lap times. A negative change from baseline indicated a better outcome.
Time Frame: Baseline (Day 1) and end of Main Portion (Week 8)
Population: The ITT Population with no missing observations at Baseline and Week 8. The test was also only performed in participants who were ambulatory.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 10 | 10
seconds | -0.712 (0.789) | -1.401 (0.788)
Statistical Analysis 1: Comparison: Placebo vs Zilucoplan 0.3 mg/kg; Test type: Superiority; p = 0.496, Linear Mixed Effect Model — Based on a linear model with treatment and strata (anti-3-hydroxy-3-methyl-glutaryl-coenzyme A reductase [HMGCR]+/anti-signal recognition particle [SRP]+) as fixed factors with Baseline 3TUG as a covariate; Least squares (LS) mean difference = -0.688, 95% CI 2-sided [-2.781 to 1.404] — The difference presented is zilucoplan 0.3 mg/kg minus placebo

5. Secondary Outcome: Change From Baseline to Week 8 in Proximal Manual Muscle Testing (MMT) Score
Description: The proximal MMT assessed muscle strength using manual muscle testing in 7 muscle groups (left and right sides assessed separately). The total MMT score for this study, inclusive of both sides, could range from 0-140, where 0 means no strength in any muscles and 140 means full strength in all the muscles examined. A negative change from Baseline indicated a worse outcome.
Time Frame: Baseline (Day 1) and end of Main Portion (Week 8)
Population: The ITT Population with no missing observations at Baseline and Week 8.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 14 | 11
score on a scale | -0.18 (3.44) | 3.71 (3.81)
Statistical Analysis 1: Comparison: Placebo vs Zilucoplan 0.3 mg/kg; Test type: Superiority; p = 0.431, Linear Mixed Effect Model — Based on a linear model with treatment and strata (anti-HMGCR+/anti-SRP+) as fixed factors with Baseline proximal MMT as a covariate; LS mean difference = 3.89, 95% CI 2-sided [-6.18 to 13.95] — The difference presented is zilucoplan 0.3 mg/kg minus placebo

6. Secondary Outcome: Change From Baseline to Week 8 in Physician Global Activity Visual Analogue Scale (VAS) Score
Description: The Physician Global Activity VAS Score measured the treating physician's global evaluation of the participant's overall disease activity using a 10 cm VAS labelled with "no activity" at the left end and "maximum activity" at the right end. The Physician Global Activity VAS Score ranged from 0 (absent extramuscular disease activity) to 10 (maximum extramuscular disease activity). A negative change from Baseline indicated a better outcome.
Time Frame: Baseline (Day 1) and end of Main Portion (Week 8)
Population: The ITT Population with no missing observations at Baseline and Week 8.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 15 | 11
score on a scale | -0.626 (0.557) | -0.830 (0.671)
Statistical Analysis 1: Comparison: Placebo vs Zilucoplan 0.3 mg/kg; Test type: Superiority; p = 0.800, Linear Mixed Effect Model — Based on a linear model with treatment and strata (anti-HMGCR+/anti-SRP+) as fixed factors with Baseline Physician Global Activity VAS as a covariate; LS mean difference = -0.204, 95% CI 2-sided [-1.855 to 1.448] — The difference presented is zilucoplan 0.3 mg/kg minus placebo

7. Secondary Outcome: Change From Baseline to Week 8 in Patient Global Activity VAS Score
Description: The Patient Global Activity VAS Score measured the treating participant's global evaluation of their overall disease activity using a 10 cm VAS labelled with "no activity" at the left end and "maximum activity" at the right end. The Patient Global Activity VAS score ranged from 0 (absent extramuscular disease activity) to 10 (maximum extramuscular disease activity). A negative change from Baseline indicated a better outcome.
Time Frame: Baseline (Day 1) and end of Main Portion (Week 8)
Population: The ITT Population with no missing observations at Baseline and Week 8.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 15 | 11
score on a scale | -0.685 (0.707) | -1.966 (0.854)
Statistical Analysis 1: Comparison: Placebo vs Zilucoplan 0.3 mg/kg; Test type: Superiority; p = 0.221, Linear Mixed Effect Model — Based on a linear model with treatment and strata (anti-HMGCR+/anti-SRP+) as fixed factors with Baseline Patient Global Activity VAS as a covariate; LS mean difference = -1.281, 95% CI 2-sided [-3.390 to 0.829] — The difference presented is zilucoplan 0.3 mg/kg minus placebo

8. Secondary Outcome: Change From Baseline to Week 8 in HAQ Score
Description: The HAQ had 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities with 2 to 3 questions for each section. Scoring within each section ranged from 0 (without any difficulty) to 3 (unable to do). The total HAQ score was then calculated by summing the scores and dividing by the number of categories answered. The total HAQ score for this study could range from 0-3, where 0 means no functional impairment and 3 means complete functional impairment. A negative change from Baseline indicated a better outcome.
Time Frame: Baseline (Day 1) and end of Main Portion (Week 8)
Population: The ITT Population with no missing observations at Baseline and Week 8.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 15 | 11
score on a scale | 0.022 (0.151) | -0.125 (0.183)
Statistical Analysis 1: Comparison: Placebo vs Zilucoplan 0.3 mg/kg; Test type: Superiority; p = 0.508, Linear Mixed Effect Model — Based on a linear model with treatment and strata (anti-HMGCR+/anti-SRP+) as fixed factors with Baseline HAQ as a covariate; LS mean difference = -0.147, 95% CI 2-sided [-0.601 to 0.307] — The difference presented is zilucoplan 0.3 mg/kg minus placebo

9. Secondary Outcome: Change From Baseline to Week 8 in MDAAT Extramuscular Disease Activity VAS Score
Description: The MDAAT extramuscular disease activity VAS score measured the degree of disease activity of extramuscular organ systems and muscle. The scoring was performed by the physician and ranged from 0 (absent extramuscular disease activity) to 10 (maximum extramuscular disease activity). A negative change from Baseline indicated a better outcome.
Time Frame: Baseline (Day 1) and end of Main Portion (Week 8)
Population: The ITT Population with no missing observations at Baseline and Week 8.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 15 | 11
score on a scale | -0.144 (0.336) | -0.287 (0.398)
Statistical Analysis 1: Comparison: Placebo vs Zilucoplan 0.3 mg/kg; Test type: Superiority; p = 0.765, Linear Mixed Effect Model; Based on a linear model with treatment and strata (anti-HMGCR+/anti-SRP+) as fixed factors with Baseline MDAAT as a covariate; LS mean difference = -0.143, 95% CI 2-sided [-1.123 to 0.837] — The difference presented is zilucoplan 0.3 mg/kg minus placebo

10. Secondary Outcome: Change From Baseline to Week 8 in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale Score
Description: The FACIT-Fatigue Scale is a 13-item tool which measured an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue was measured on a 4-point Likert scale. The total FACIT-Fatigue Scale score for this study could range from 0-52, where 0 means the participants were very much fatigued during their usual daily activities and 52 means the participants were not at all fatigued during their usual daily activities. A negative change from Baseline indicated a worse outcome.
Time Frame: Baseline (Day 1) and end of Main Portion (Week 8)
Population: The ITT Population with no missing observations at Baseline and Week 8.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Zilucoplan 0.3 mg/kg
Number analyzed (Participants) | 15 | 11
score on a scale | 3.45 (3.41) | 8.98 (4.08)
Statistical Analysis 1: Comparison: Placebo vs Zilucoplan 0.3 mg/kg; Test type: Superiority; p = 0.265, Linear Mixed Effect Model — Based on a linear model with treatment and strata (anti-HMGCR+/anti-SRP+) as fixed factors with Baseline FACIT-Fatigue Scale as a covariate; LS mean difference = 5.53, 95% CI 2-sided [-4.49 to 15.55] — The difference presented is zilucoplan 0.3 mg/kg minus placebo

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) to End of Safety Follow-up (Week 83)
Description: The Safety Population included all participants who have received at least 1 dose of study drug, with participants analyzed based on the actual study treatment received.
Groups:
- Extension Portion: Zilucoplan 0.3 mg/kg: Participants received daily SC doses of zilucoplan 0.3 mg/kg during the Extension Portion of the study.
Arm/Group | Main Portion: Placebo | Main Portion: Zilucoplan 0.3 mg/kg | Extension Portion: Zilucoplan 0.3 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/12 | 1/25
Serious Adverse Events (participants affected / at risk) | 3/15 | 0/12 | 8/25
Other Adverse Events (participants affected / at risk) | 13/15 | 9/12 | 15/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Portion: Placebo (N=15) | Main Portion: Zilucoplan 0.3 mg/kg (N=12) | Extension Portion: Zilucoplan 0.3 mg/kg (N=25)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 3 (4)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Portion: Placebo (N=15) | Main Portion: Zilucoplan 0.3 mg/kg (N=12) | Extension Portion: Zilucoplan 0.3 mg/kg (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 1 (1) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 1 (2) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 4 (4) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated based on the primary efficacy endpoint analysis after the first data lock.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/32/NCT04025632/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/32/NCT04025632/SAP_001.pdf